CLINICAL TRIAL: NCT06492252
Title: Sensorimotor Basis of Speech Motor Learning and Retention
Brief Title: Speech Motor Learning and Retention (Aim 3)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000037622_c; 1R01DC022097-01A1 (NIH)
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Speech
Keywords: Speech Motor Learning; Retention
MeSH Terms: conditions — Speech | interventions — Magnetic Resonance Imaging; Acclimatization

STUDY DESIGN:
Intervention Model Description: Healthy right-handed adults with normal hearing will be recruited in equal number from both sexes. All participants will be fluent English speakers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Altered auditory feedback + fMRI (Experimental): Participants will perform learning tasks then undergo fMRI. This procedure will be repeated on day 2. Functional connectivity patterns between regions that predict learning will be assessed. Participants then leave the laboratory and return 24 hours later to assess retention of learning.
  Interventions: Device: fMRI; Behavioral: Adaptation
- Control Condition (Experimental): Participants in a control condition who will undergo the same procedures, without altered feedback
  Interventions: Device: fMRI; Behavioral: Adaptation

INTERVENTIONS:
Device: fMRI — To assess functional connectivity patterns between regions that predict learning.
Behavioral: Adaptation — Auditory adaptation in speech
  Arms: Altered auditory feedback + fMRI
Behavioral: Adaptation — Auditory baseline in speech
  Arms: Control Condition

SUMMARY:
The overall goal of this research is to test a new model of speech motor learning, whose central hypothesis is that learning and retention are associated with plasticity not only in motor areas of the brain but in auditory and somatosensory regions as well. The strategy for the proposed research is to identify individual brain areas that contribute causally to retention by disrupting their activity with transcranial magnetic stimulation (TMS). Investigators will also use functional magnetic resonance imaging (fMRI) which will enable identification of circuit-level activity which predicts either learning or retention of new movements, and hence test the specific contributions of candidate sensory and motor zones. In other studies, investigators will record sensory and motor evoked potentials over the course of learning to determine the temporal order in which individual sensory and cortical motor regions contribute. The goal here is to identify brain areas in which learning-related plasticity occurs first and which among these areas predict subsequent learning.

DETAILED DESCRIPTION:
The focus of this registration is Aim 3. Excitability will be assessed. In Aim 3, resting-state fMRI will be interleaved with speech motor adaptation, again using Harvard Sentences. Additional scans and retention tests will be conducted 24 hours later, to assess motor memory consolidation.

The Speech Motor Learning and Retention Master Protocol is NCT06467292.

ELIGIBILITY:
Inclusion Criteria:

* Fluent English speakers
* Right-handed
* Normal hearing
* No speech disorder or reading disability

Exclusion Criteria:

* Cardiac pacemaker
* Aneurysm clip
* Heart or Vascular clip
* Prosthetic valve
* Metal implants
* Metal in brain, skull, or spinal cord
* Implanted neurostimulator
* Medication infusion device
* Cochlear implant or tinnitus (ringing in ears)
* Personal and/or family history of epilepsy or other neurological disorders or history of head concussion
* Psychoactive medications
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Speech motor learning | Performance as measured at the end of learning (30 minute session)
  Audapter software will be used to alter the first and second formant frequencies of the spoken words and this is played back to subjects through headphones. Subjects will be tested both with unaltered feedback and with abruptly introduced frequency shifts.The change in the first (F1) and second format frequency (F2) values will be assessed using Praat.
Retention of learning | 24 hours after learning (re-test lasts 30 minutes)
  The retention of adaptation to altered auditory feedback (and relearning) will be quantified in terms of F1 and F2 frequency shifts (relative to pre-training baseline). Larger values indicate more complete relearning or retention.
Change in fMRI resting-state connectivity following speech motor learning | baseline and at the end of learning (30 minute session)
  fMRI resting-state connectivity change following speech motor learning. Functional connectivity will be measured between each of the following regions: Heschel's gyrus, posterior superior temporal gyrus, primary and second somatosensory cortex, supramarginal gyrus, inferior frontal gyrus, motor and ventral premotor cortex and supplementary motor area.
fMRI resting-state connectivity measures of motor memory retention | 24 hours after learning (re-test lasts 30 minutes)
  fMRI resting-state connectivity measures of motor memory retention. Functional connectivity will be measured between each of the following regions: Heschel's gyrus, posterior superior temporal gyrus, primary and second somatosensory cortex, supramarginal gyrus, inferior frontal gyrus, motor and ventral premotor cortex and supplementary motor area.

CONTACTS AND LOCATIONS:
Overall Officials: David Ostry, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No